CLINICAL TRIAL: NCT04115293
Title: A Phase 3, Multicenter, Randomized, Double Blind, Placebo-Controlled Study to Confirm the Safety, Tolerability, and Efficacy of Zilucoplan in Subjects With Generalized Myasthenia Gravis
Brief Title: Safety, Tolerability, and Efficacy of Zilucoplan in Subjects With Generalized Myasthenia Gravis
Acronym: RAISE
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Ra Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Organization: UCB Pharma (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: RA101495-02.301
Record Dates: First submitted 2019-10-02; First posted 2019-10-04 (Actual); Results first posted 2023-01-17 (Actual); Last update posted 2025-07-16 (Actual); Status verified 2025-07

CONDITIONS: Myasthenia Gravis, Generalized
MeSH Terms: conditions — Myasthenia Gravis | interventions — zilucoplan

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- 0.3 mg/kg zilucoplan (RA101495) (Experimental)
  Interventions: Drug: zilucoplan (RA101495)
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: zilucoplan (RA101495) — Daily subcutaneous (SC) injection
  Arms: 0.3 mg/kg zilucoplan (RA101495)
Drug: Placebo — Daily subcutaneous (SC) injection
  Arms: Placebo

SUMMARY:
The RAISE study is a multicenter, randomized, double-blind, placebo controlled study to confirm the efficacy, safety, and tolerability of zilucoplan in subjects with generalized Myasthenia Gravis. Subjects will be randomized in a 1:1 ratio to receive daily SC doses of 0.3 mg/kg zilucoplan or placebo for 12 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of gMG [Myasthenia Gravis Foundation of America (MGFA) Class II-IV] at Screening
* Positive serology for acetylcholine receptor (AChR) autoantibodies
* MG-ADL Score of ≥ 6 at Screening and Baseline
* QMG score ≥ 12 at Screening and Baseline
* No change in corticosteroid dose for at least 30 days prior to Baseline or anticipated to occur during the 12-week Treatment Period
* No change in immunosuppressive therapy, including dose, for at least 30 days prior to Baseline or anticipated to occur during the 12-week Treatment Period

Exclusion Criteria:

* Thymectomy within 12 months prior to Baseline or scheduled to occur during the 12 week Treatment Period
* History of meningococcal disease
* Current or recent systemic infection within 2 weeks prior to Baseline or injection requiring intravenous (IV) antibiotics within 4 weeks prior to Baseline

Ages: 18 Years to 74 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 174 (Actual)
Dates: Start 2019-09-17 (Actual); Primary Completion 2021-12-30 (Actual); Study Completion 2021-12-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: UCB Cares, Study Director — 0018445992273 (UCB)
Locations (77):
- United States (37):
  - Site 41: Diagnostic and Medical Clinic, Mobile, Alabama
  - Site 116: Neuromuscular Clinic and Research Center, Phoenix, Arizona
  - Site 4: University of Southern California, Los Angeles, California
  - Site 31: University of California Irvine, Orange, California
  - Site 220: Investigator Site, Pasadena, California
  - Site 160: Forbes Norris MDA/ALS Research and Treatment Center, San Francisco, California
  - Site 24: Yale University, New Haven, Connecticut
  - Site 27: George Washington University, Washington D.C., District of Columbia
  - Site 182: Gelasio Baras Neurology, Miami, Florida
  - Site 25: University of South Florida, Tampa, Florida
  - Site 135: Augusta University Medical Center, Augusta, Georgia
  - Site 176: Hawaii Pacific Neuroscience, Honolulu, Hawaii
  - Site 188: North Shore Medical Group - Glenview, Glenview, Illinois
  - Site 156: Indiana University Health Neuroscience Center, Indianapolis, Indiana
  - Site 32: Kansas University Medical Center Research Institute, Kansas City, Kansas
  - Site 221: Neurology Center of New England, Foxborough, Massachusetts
  - Site 33: Detroit medical Center - University Health Center, Detroit, Michigan
  - Site 49: Michigan State University, East Lansing, Michigan
  - Site 127: University of Minnesota, Minneapolis, Minnesota
  - Site 134: Neurology and Sleep Disorders Clinic, Columbia, Missouri
  - Site 117: Las Vegas Clinic, Las Vegas, Nevada
  - Site 123: Northwell Health Neuroscience Institute, Great Neck, New York
  - Site 23: Hospital for Special Surgery, New York, New York
  - Site 47: Mount Sinai Hospital, New York, New York
  - Site 22: University of North Carolina, Chapel Hill, North Carolina
  - Site 15: Duke University, Durham, North Carolina
  - Site 122: Cleveland Clinic, Cleveland, Ohio
  - Site 38: Ohio State University, Columbus, Ohio
  - Site 40: Allegheny Neurological Associates, Pittsburgh, Pennsylvania
  - Site 128: Medical University of South Carolina, Charleston, South Carolina
  - Site 185: Neurology Clinic Cordova, Cordova, Tennessee
  - Site 131: Austin Neuromuscular Center, Austin, Texas
  - Site 19: University of Texas Southwestern, Dallas, Texas
  - Site 39: University of Utah, Salt Lake City, Utah
  - Site 164: University of Virginia Health System, Charlottesville, Virginia
  - Site 154: University of Washington, Seattle, Washington
  - Site 45: Center for Neurological Disorders, Milwaukee, Wisconsin
- Canada (2):
  - Site 44: London Health Sciences Centre University Hospital, London, Ontario
  - Site 11: Montreal Neurological Institute and Hospital (McGill University), Montreal, Quebec
- France (5):
  - Site 191: Centre Hosptitalier Universitaire d'Angers, Angers
  - Site 204: Centre Hospitalier Régional Universitaire de Lille, Lille
  - Site 118: Hôpital Pasteur, Nice
  - Site 105: Pitié-Salpêtrière University Hospital, Paris
  - Site 137: Les Hôpitaux Universitaires de Strasbourg, Strasbourg
- Germany (2):
  - Site 150: Universitätsmedizin Göttingen, Göttingen
  - Site 129: Universitätsklinikum Tübingen, Tübingen
- Italy (2):
  - Site 126: Fondazione IRCCS Istituto Neurologico Carlo Besta, Milan
  - Site 132: Università Cattolica del Sacro Cuore - Campus di Milano, Roma
- Japan (11):
  - Site 169: International University of Health and Welfare Narita Hospital, Narita, Chiba
  - Site 151: Chiba University Hospital, Chiba
  - Site 136: General Hanamaki Hospital, Iwata
  - Site 179: Kagawa University Hospital - Collagen disease/Rheumatic int, Kita-gun
  - Site 146: Nagasaki University Hospital, Nagasaki
  - Site 152: Hokkaido Medical Center, Sapporo
  - Site 144: Sendai Medical Center, Sendai
  - Site 153: Toho University Ohashi Medical Center, Tokyo
  - Site 163: Tokyo Medical University Hospital, Tokyo
  - Site 141: Keio University Hospital, Tokyo
  - Site 165: Osaka University Hospital, Tokyo
- Norway (2):
  - Site 140: Haukeland University Hospital / Health Bergen, Bergen
  - Site 143: Oslo Universitetssykehus, Oslo
- Poland (11):
  - Site 209: Niepubliczny Zakład Opieki Zdrowotnej NEURO - KARD, Poznan, Greater Poland Voivodeship
  - Site 192: Krakowski Szpital Specjalistyczny im. Jana Pawła II, Krakow, Lesser Poland Voivodeship
  - Site 205: Prywatny Gabinet Lekarski Urszula Chyrchel-Paszkiewicz, Lublin, Lublin Voivodeship
  - Site 194: Twoja Przychodnia - Centrum Medyczne Nowa Sól, Nowa Sól, Lubusz Voivodeship
  - Site 214: AmiCare Centrum Medyczne, Lodz, Lódzkie
  - Site 201: Centrum Medyczne Pratia - Warszawa, Warsaw, Masovian Voivodeship
  - Site 195: Wielospecjalistyczna Poradnia Lekarska Synapsis, Katowice, Silesian Voivodeship
  - Site 213: Niepubliczny Zakład Opieki Zdrowotnej NOVO-MED, Katowice, Silesian Voivodeship
  - Site 193: Krakowska Akademia Neurologii - Centrum Neurologii Kliniczne, Krakow
  - Site 211: Specjalistyczne Gabinety Sp. z o.o., Krakow
  - Site 210: Clinhouse Centrum Medyczne, Lublin
- Spain (3):
  - Site 133: Hospital Universitari Vall d'Hebrón, Barcelona
  - Site 168: Hospital de la Santa Creu i Sant Pau, Barcelona
  - Site 138: Hospital Universitario de Basurto, Bilbao
- United Kingdom (2):
  - Site 119: Oxford University Hospitals NHS Foundation Trust, Oxford
  - Site 130: Royal Hallamshire Hospital, Sheffield

IPD SHARING:
Plan to Share IPD: Yes
Data from this trial may be requested by qualified researchers six months after product approval in the US and/or Europe, or global development is discontinued, and 18 months after trial completion. Investigators may request access to anonymized individual patient-level data and redacted trial documents which may include: analysis-ready datasets, study protocol, annotated case report form, statistical analysis plan, dataset specifications, and clinical study report. Prior to use of the data, proposals need to be approved by an independent review panel at www.Vivli.org and a signed data sharing agreement will need to be executed. All documents are available in English only, for a prespecified time, typically 12 months, on a password protected portal. This plan may change if the risk of re-identifying trial participants is determined to be too high after the trial is completed;in this case and to protect participants, individual patient-level data would not be made available.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Data from this trial may be requested by qualified researchers six months after product approval in the US and/or Europe or global development is discontinued, and 18 months after trial completion.
Access Criteria: Qualified researchers may request access to anonymized IPD and redacted study documents which may include: raw datasets, analysis-ready datasets, study protocol, blank case report form, annotated case report form, statistical analysis plan, dataset specifications, and clinical study report. Prior to use of the data, proposals need to be approved by an independent review panel at www.Vivli.org and a signed data sharing agreement will need to be executed. All documents are available in English only, for a pre-specified time, typically 12 months, on a password protected portal.
URL: http://www.Vivli.org

REFERENCES:
- [Result] Howard JF Jr, Bresch S, Genge A, Hewamadduma C, Hinton J, Hussain Y, Juntas-Morales R, Kaminski HJ, Maniaol A, Mantegazza R, Masuda M, Sivakumar K, Smilowski M, Utsugisawa K, Vu T, Weiss MD, Zajda M, Boroojerdi B, Brock M, de la Borderie G, Duda PW, Lowcock R, Vanderkelen M, Leite MI; RAISE Study Team. Safety and efficacy of zilucoplan in patients with generalised myasthenia gravis (RAISE): a randomised, double-blind, placebo-controlled, phase 3 study. Lancet Neurol. 2023 May;22(5):395-406. doi: 10.1016/S1474-4422(23)00080-7. PMID 37059508
- [Result] Weiss MD, Freimer M, Leite MI, Maniaol A, Utsugisawa K, Bloemers J, Boroojerdi B, Howard E, Savic N, Howard JF Jr. Improvement of fatigue in generalised myasthenia gravis with zilucoplan. J Neurol. 2024 May;271(5):2758-2767. doi: 10.1007/s00415-024-12209-3. Epub 2024 Feb 24. PMID 38400914
- [Result] de la Borderie G, Chimits D, Boroojerdi B, Brock M, Duda PW, Grimson F, Mahoney P, Strimenopoulou F, Cutter G, Aban I, Brauner S, Petersson M, Howard JF Jr, Bennett N. Maintenance of zilucoplan efficacy in patients with generalised myasthenia gravis up to 24 weeks: a model-informed analysis. Ther Adv Neurol Disord. 2024 Sep 21;17:17562864241279125. doi: 10.1177/17562864241279125. eCollection 2024. PMID 39314260
- [Result] Hewamadduma C, Freimer M, Genge A, Leite MI, Utsugisawa K, Vu T, Boroojerdi B, Grimson F, Savic N, Vanderkelen M, Howard JF Jr; RAISE-XT study team. Changes in corticosteroid and non-steroidal immunosuppressive therapy with long-term zilucoplan treatment in generalized myasthenia gravis. J Neurol. 2025 Jun 12;272(7):457. doi: 10.1007/s00415-025-13113-0. PMID 40504283

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study started to enroll participants in September 2019 and concluded in December 2021.
Pre-assignment Details: The Participant flow refers to the Randomized Set.
Groups:
- Placebo: Participants self-administered zilucoplan (RA101495) matching placebo as subcutaneous (SC) injection during 12-week Treatment Period.
- Zilucoplan 0.3 mg/kg: Participants self-administered zilucoplan (RA101495) 0.3 milligrams/kilogram/day (mg/kg/day) SC injection during 12-week Treatment Period.
Period: Overall Study
Arm/Group | Placebo | Zilucoplan 0.3 mg/kg
Started | 88 | 86
Completed | 84 | 82
Not Completed | 4 | 4
Not completed — Adverse Event | 0 | 2
Not completed — Withdrawal by Subject | 2 | 1
Not completed — Physician Decision | 1 | 0
Not completed — Death | 1 | 1

BASELINE CHARACTERISTICS:
Population: The modified Intention-to-Treat (mITT) population included all randomized participants who received at least 1 dose of study drug and had at least 1 post-dosing MG-ADL score.
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Zilucoplan 0.3 mg/kg | Total
Number analyzed (Participants) | 88 | 86 | 174
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 62 | 64 | 126
  >=65 years | 26 | 22 | 48
Age, Continuous [Mean (Standard Deviation); unit: years] | 53.3 (15.7) | 52.6 (14.6) | 53.0 (15.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 47 | 52 | 99
  Male | 41 | 34 | 75
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  American Indian/Alaska native | 1 | 0 | 1
  Asian | 14 | 7 | 21
  Black | 7 | 6 | 13
  Native Hawaiian or other Pacific Islander | 0 | 0 | 0
  White | 62 | 66 | 128
  Other/Mixed | 0 | 0 | 0
  Missing | 4 | 7 | 11
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Hispanic or Latino | 5 | 7 | 12
  Not Hispanic or Latino | 79 | 72 | 151
  Missing | 4 | 7 | 11

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline (CFB) to Week 12 in Myasthenia Gravis-Activities of Daily Living (MG-ADL) Total Score
Description: The MG-ADL is an 8-item patient-reported outcome measure assessing MG symptoms and their effects on daily activities. Each item in the scale scored 0 to 3 (0=None, 3=severe disease) point scale. The total score was the sum of all individual item scores and ranged from 0 to 24. Higher scores indicated more severe disability due to MG. A decrease from Baseline score indicated improvement.
Time Frame: From Baseline to End of Treatment (Week 12)
Population: as for baseline characteristics
Measure: Least Squares Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Placebo | Zilucoplan 0.3 mg/kg
Number analyzed (Participants) | 88 | 86
score on a scale | -2.30 [-3.17 to -1.43] | -4.39 [-5.28 to -3.50]
Statistical Analysis 1: Comparison: Placebo vs Zilucoplan 0.3 mg/kg; Test type: Superiority; p < 0.001, MMRM ANCOVA; LS Mean Difference = -2.09, 95% CI 2-sided [-3.24 to -0.95]

2. Secondary Outcome: Change From Baseline to Week 12 in the Quantitative Myasthenia Gravis (QMG) Total Score
Description: The QMG is a standardized and validated quantitative strength scoring system that was developed specifically for MG. The scale consisted of 13 items. Each item in the scale scored on a 0 to 3-point scale, ranging from 0 (no weakness) to 3 (severe weakness), summing up to the overall score range from 0 to 39. Higher scores indicated more severe impairment. A decrease from Baseline score indicated improvement.
Time Frame: From Baseline to End of Treatment (Week 12)
Population: as for baseline characteristics
Measure: Least Squares Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Placebo | Zilucoplan 0.3 mg/kg
Number analyzed (Participants) | 88 | 86
score on a scale | -3.25 [-4.32 to -2.17] | -6.19 [-7.29 to -5.08]
Statistical Analysis 1: Comparison: Placebo vs Zilucoplan 0.3 mg/kg; Test type: Superiority; p < 0.001, MMRM ANCOVA; LS Mean Difference = -2.94, 95% CI 2-sided [-4.39 to -1.49]

3. Secondary Outcome: Change From Baseline to Week 12 in the Myasthenia Gravis Composite (MGC) Scale Total Score
Description: The total MGC score was sum of responses to 10 individual items : 1. Ptosis upward gaze (0 to 3), 2. Double vision on lateral gaze, left or right (0, to 4), 3. Eye closure (0 to 2), 4. Talking (0 to 6), 5. Chewing (0 to 6), 6. Swallowing [0 to 6], 7. Breathing (0 to 9), 8. Neck flexion or extension (0 to 4), 9. Shoulder abduction (0 to 5), 10. Hip flexion (0 to 5). The higher score for each item indicated severity. The total score ranged 0 to 50 with higher score indicative of severe disease activity). A decrease from Baseline score showed improvement.
Time Frame: From Baseline to End of Treatment (Week 12)
Population: as for baseline characteristics
Measure: Least Squares Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Placebo | Zilucoplan 0.3 mg/kg
Number analyzed (Participants) | 88 | 86
score on a scale | -5.42 [-6.98 to -3.86] | -8.62 [-10.22 to -7.01]
Statistical Analysis 1: Comparison: Placebo vs Zilucoplan 0.3 mg/kg; Test type: Superiority; p = 0.0023, MMRM ANCOVA; LS Mean Difference = -3.20, 95% CI 2-sided [-5.24 to -1.16]

4. Secondary Outcome: Change From Baseline to Week 12 in the Myasthenia Gravis - Quality of Life Revised (MG-QoL15r) Scale Total Score
Description: The MG-QoL15r is a 15-item patient-reported outcome measure designed to assess quality of life in patients with MG. Each item in the scale scored on a 0 to 2-point scale (0=Not much at all, 1=Somewhat, 2=Very much). The total score was the sum of the 15 individual item scores, ranging from 0 to 30. Higher scores indicated more severe impact of the disease on aspects of the patient's life. A decrease from Baseline score indicated improvement.
Time Frame: From Baseline to End of Treatment (Week 12)
Population: as for baseline characteristics
Measure: Least Squares Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Placebo | Zilucoplan 0.3 mg/kg
Number analyzed (Participants) | 88 | 86
score on a scale | -3.16 [-4.65 to -1.67] | -5.65 [-7.17 to -4.12]
Statistical Analysis 1: Comparison: Placebo vs Zilucoplan 0.3 mg/kg; Test type: Superiority; p = 0.0128, MMRM ANCOVA; LS Mean Difference = -2.49, 95% CI 2-sided [-4.45 to -0.54]

5. Secondary Outcome: Time to First Receipt of Rescue Therapy Over the 12-week Treatment Period
Description: Time to first receipt of rescue therapy over the 12-week treatment period (in days) was defined as the date of first rescue therapy use minus date of first Investigational Medicinal Product (IMP) + 1.
Time Frame: From Baseline to End of Treatment (Week 12)
Population: as for baseline characteristics
Measure: Median (Full Range); unit: Days
Arm/Group | Placebo | Zilucoplan 0.3 mg/kg
Number analyzed (Participants) | 88 | 86
Days | NA [NA to NA] — The median time to first receipt of rescue therapy was not estimated due to the less number of events. | NA [NA to NA] — The median time to first receipt of rescue therapy was not estimated due to the less number of events.

6. Secondary Outcome: Percentage of Participants Achieving Minimal Symptom Expression (MSE) at Week 12 Without Rescue Therapy
Description: Percentage of Participants achieving MSE was defined as achieving a MG-ADL value of a 0 (No MG symptoms) or 1 (Mild MG symptoms) at Week 12 and not having taken rescue therapy. Any participant with an event of death, myasthenic crisis or rescue therapy was considered as non-responders. Any other missing data was imputed using the missing at Random (MAR) assumption.
Time Frame: End of Treatment (Week 12)
Population: The mITT population included randomized participants who received at least 1 dose of study drug and had at least 1 post-dosing MG-ADL score.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Zilucoplan 0.3 mg/kg
Number analyzed (Participants) | 88 | 86
percentage of participants | 5.8 | 14.0
Statistical Analysis 1: Comparison: Placebo vs Zilucoplan 0.3 mg/kg; Test type: Superiority; p = 0.0885, Regression, Logistic; Odds Ratio (OR) = 2.608, 95% CI 2-sided [0.866 to 7.860]

7. Secondary Outcome: Percentage of Participants Achieving a ≥ 3-point Reduction in MG-ADL Score at Week 12 Without Rescue Therapy
Description: Percentage of participants achieving a ≥ 3-point reduction in MG-ADL Score at Week 12 without rescue therapy were reported. The MG-ADL is an 8-item patient-reported outcome measure assessing MG symptoms and their effects on daily activities. Each item in the scale scored on a 0 to 3 (0=None, 3=severe disease) point scale. The total score was the sum of all individual item scores and ranged from 0 to 24. Higher scores indicated more severe disability due to MG. Any participant with an event of death, myasthenic crisis or rescue therapy was considered as non-responders. Any other missing data was imputed using the MAR assumption.
Time Frame: End of Treatment (Week 12)
Population: as for outcome 6
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Zilucoplan 0.3 mg/kg
Number analyzed (Participants) | 88 | 86
percentage of participants | 46.1 | 73.1
Statistical Analysis 1: Comparison: Placebo vs Zilucoplan 0.3 mg/kg; Test type: Superiority; p < 0.001, Regression, Logistic; Odds Ratio (OR) = 3.184, 95% CI 2-sided [1.662 to 6.101]

8. Secondary Outcome: Percentage of Participants Achieving a ≥5-point Reduction in QMG Score Without Rescue Therapy at Week 12
Description: Percentage of participants achieving a ≥5-point reduction in QMG Score without rescue therapy at Week 12 were reported. The QMG is a standardized and validated quantitative strength scoring system that was developed specifically for MG. The scale consisted of 13 items. Each item in the scale scored on a 0 to 3-point scale, ranging from 0 (no weakness) to 3 (severe weakness), summing up to the overall score range from 0 to 39. Higher scores indicated more severe impairment. Any participant with an event of death, myasthenic crisis or rescue therapy was considered as non-responders. Any other missing data was imputed using the MAR assumption.
Time Frame: End of Treatment (Week 12)
Population: as for outcome 6
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Zilucoplan 0.3 mg/kg
Number analyzed (Participants) | 88 | 86
percentage of participants | 33.0 | 58.0
Statistical Analysis 1: Comparison: Placebo vs Zilucoplan 0.3 mg/kg; Test type: Superiority; p = 0.0012, Regression, Logistic; Odds Ratio (OR) = 2.865, 95% CI 2-sided [1.518 to 5.409]

9. Secondary Outcome: Percentage of Participants With Treatment-emergent Adverse Events (TEAEs)
Description: A TEAE is defined as an AE starting on or after the time of first administration of IMP and up to and including 40 days after the final dose (or last contact depending on which occurs first). Adverse events starting before the date of the first administration of IMP were not considered TEAEs.
Time Frame: From Baseline (Day 1) to Safety Follow-up visit (19 Weeks [12 weeks Treatment Period plus up to 7 weeks Follow-up])
Population: The Safety Set (SS) included all participants who received at least 1 dose of study drug based on the actual study treatment received.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Zilucoplan 0.3 mg/kg
Number analyzed (Participants) | 88 | 86
percentage of participants | 70.5 | 76.7

ADVERSE EVENTS:
Time Frame: From Baseline (Day 1) to Safety follow-up visit (19 Weeks [12 weeks Treatment Period plus up to 7 weeks follow-up])
Description: A TEAE is defined as an AE starting on or after the time of first administration of IMP and up to and including 40 days after the final dose (or last contact depending on which occurs first). Adverse events starting before the date of the first administration of IMP were not considered TEAEs.
Arm/Group | Placebo | Zilucoplan 0.3 mg/kg
All-Cause Mortality (participants affected / at risk) | 1/88 | 1/86
Serious Adverse Events (participants affected / at risk) | 13/88 | 11/86
Other Adverse Events (participants affected / at risk) | 34/88 | 41/86
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=88) | Zilucoplan 0.3 mg/kg (N=86)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (1) | 0 (0)
Aphthous ulcer (Gastrointestinal disorders) | 0 (0) | 1 (1)
Oesophageal candidiasis (Infections and infestations) | 0 (0) | 1 (1)
Oral candidiasis (Infections and infestations) | 0 (0) | 1 (1)
COVID-19 (Infections and infestations) | 2 (2) | 1 (1)
COVID-19 pneumonia (Infections and infestations) | 2 (2) | 1 (1)
Herpes simplex meningoencephalitis (Infections and infestations) | 1 (2) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 1 (1)
Sepsis (Infections and infestations) | 0 (0) | 1 (1)
Lipase increased (Investigations) | 0 (0) | 1 (1)
Metastases to meninges (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Cerebral haemorrhage (Nervous system disorders) | 1 (1) | 0 (0)
Cerebrovascular accident (Nervous system disorders) | 1 (1) | 0 (0)
Myasthenia gravis (Nervous system disorders) | 5 (6) | 2 (3)
Hyperemesis gravidarum (Pregnancy, puerperium and perinatal conditions) | 1 (1) | 0 (0)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Angioedema (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=88) | Zilucoplan 0.3 mg/kg (N=86)
Diarrhoea (Gastrointestinal disorders) | 2 (2) | 9 (9)
Vomiting (Gastrointestinal disorders) | 5 (5) | 3 (3)
Injection site bruising (General disorders) | 8 (11) | 14 (18)
Injection site pain (General disorders) | 3 (3) | 8 (9)
Urinary tract infection (Infections and infestations) | 4 (4) | 7 (7)
Nasopharyngitis (Infections and infestations) | 3 (3) | 5 (5)
Contusion (Injury, poisoning and procedural complications) | 3 (3) | 7 (8)
Lipase increased (Investigations) | 1 (1) | 6 (6)
Amylase increased (Investigations) | 2 (2) | 5 (5)
Headache (Nervous system disorders) | 14 (19) | 13 (16)
Myasthenia gravis (Nervous system disorders) | 5 (6) | 8 (10)
Rash (Skin and subcutaneous tissue disorders) | 5 (9) | 3 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (2):
  • Study Protocol (2020-12-18): https://cdn.clinicaltrials.gov/large-docs/93/NCT04115293/Prot_000.pdf
  • Statistical Analysis Plan (2021-12-06): https://cdn.clinicaltrials.gov/large-docs/93/NCT04115293/SAP_001.pdf